CLINICAL TRIAL: NCT04894851
Title: A Pilot Study of Contingency Management for Hoarding Disorder
Brief Title: Contingency Management for Hoarding Disorder
Acronym: HCM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hartford Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WORD004040HI
Record Dates: First submitted 2013-11-12; First posted 2021-05-20 (Actual); Last update posted 2021-05-20 (Actual); Status verified 2021-05

CONDITIONS: Hoarding Disorder
Keywords: Hoarding Disorder; Contingency Management; Cognitive-Behavioral Therapy; Group Therapy
MeSH Terms: conditions — Hoarding Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Contingency Management (Experimental): Receives contingency payments each month based on decluttering scores
  Interventions: Behavioral: Contingency Management

INTERVENTIONS:
Behavioral: Contingency Management — Participants in the current study will receive contingencies for improvement in clutter, as measured by a trained, independent in-home rater. Ratings will be completed by after study consent, and once every month thereafter, being conducted at weeks 0, 4, 8, 12, and 16 of treatment. Participants will be reimbursed for each new 1-point reduction in CIR score, a set dollar amount per month for each CIR point reduction they maintain from baseline. Therefore, a perfectly performing patient would earn reimbursement (A CIR reduction of 8 points made in the first month and maintained throughout treatment. If a CIR score is higher than the prior month, the reinforcement schedule will reset to zero.

SUMMARY:
Aim 1: To test the efficacy of contingency management for patients with hoarding disorder (HD).

Hypothesis 1. Participants completing CM will show significant pre- to post-treatment decreases in severity of hoarding symptoms and clinician-rated impairment, and significant increases in quality of life.

Exploratory analyses will examine whether effect sizes compare with those of prior trials of cognitive-behavioral therapy (CBT) for HD conducted within our clinic, whether problem severity at follow-up is predicted by hoarding severity measured immediately after treatment completion, and whether readiness for change improves with treatment.

DETAILED DESCRIPTION:
The primary aim of the current study is a preliminary investigation of the efficacy of contingency management (CM) in the treatment of hoarding disorder (HD). CM is a highly efficacious treatment that has been used to treat issues such as substance use disorders, medication/ medical regimen nonadherence, and schizophrenia. While the current best-practice treatment for HD (cognitive behavioral therapy; CBT) is efficacious in that it results in significant symptom reduction, many patients continue to have high levels of functional impairment and distressing symptoms after treatment completion. We strongly feel that CM is able to address many of the issues that arise in the context of CBT for hoarding and we feel that the addition of CM to as CBT will result in significant pre- to post-treatment decreases in severity of hoarding symptoms and impairment, and significant increases in quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Primary Hoarding Disorder,
* currently participating in the Hoarding Disorder treatment group at the HH Anxiety Disorders Center

Exclusion Criteria:

* Not clinically appropriate for a group treatment format (i.e., active suicidality or aggressive behavior, psychosis, current physiological substance dependence, or personality issues that would be expected to substantially interfere with the group milieu; cognitively intact).
* Participants will also be excluded if they have previously completed CBT for HD.
* In addition, participants in the CM portion of the treatment will be required to live within one hour travel time of the treatment facility to allow for home visits with the independent rater.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2013-08; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Hoarding Rating Scale (HRS) | Change from week 1 (pre) to week 16 (post)
  A brief 5-item interview to rate clutter, difficulty discarding, acquisition, distress, and impairment. Each item is rated on a likert scale from 1 to 8, with higher scores reflective of higher symptom severity.
Clutter Image Rating Scale | Change from week 1 (pre) to week 16 (post)
  A pictorial measure of clutter severity containing nine photographs depicting increasing levels of clutter. CIR Scores can range from 1 to 9, with picture 1 indicating an absence of clutter and 9 indicative of the highest level of clutter. Each available room will be rated.

SECONDARY OUTCOMES:
Readiness Ruler | Change from week 1 (pre) to week 16 (post)
  The Readiness Ruler is a brief measure of motivation, which prompts patients with a 10-point likert scale on which they rate readiness, with a score of 0 reflecting "not ready," and a score of 10 reflecting "ready." The Readiness Ruler used in the current study will have patients rate both readiness for treatment and readiness for change.
The World Health Organization Quality of Life Scale (WHOQOL-BREF) | Change from week 1 (pre) to week 16 (post)
  Was developed by the World Health Organization and field-tested in 18 countries (including the United States) and contains 26 self-report questions, which measure the following broad domains: physical health, psychological health, social relationships, and environment. These four scales can be summed to calculate a total quality of life (QOL) score, ranging from 0 (least favorable health status)to 100 (most favorable health status).

CONTACTS AND LOCATIONS:
Overall Officials: Blaise L Worden, Ph.D., Principal Investigator — Hartford Hospital
Locations (1):
- Anxiety Disorders Center, Institute of Lilving, Hartford, Connecticut, United States